CLINICAL TRIAL: NCT04840511
Title: The Effect of Perioperative Lidocaine Infusion on Neutrophil Extracellular Trapping in the Patients Undergoing the Robot-assisted Prostatectomy
Brief Title: The Effect of Perioperative Lidocaine Infusion on Neutrophil Extracellular Trapping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NETosis-prostate Ca
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Urologic Cancer
MeSH Terms: conditions — Urologic Neoplasms | interventions — Lidocaine; Control Groups; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Experimental): The study group receives perioperative lidocaine infusion with general anesthesia for robot-assisted prostatectomy
  Interventions: Drug: lidocaine group
- control group (Placebo Comparator): The control group receives normal saline infusion with with general anesthesia for robot-assisted prostatectomy
  Interventions: Drug: control group

INTERVENTIONS:
Drug: lidocaine group — lidocaine 1.5 mg/kg bolus (infused over 10 min) followed by 2.0 mg/kg/h during operation and 1.0 mg/kg/h during postoperative 24 hours (no more than 120 mg/h)
  Other Names: lidocaine
  Arms: lidocaine group
Drug: control group — normal saline 0.15 ml bolus followed by 0.2 ml/kg/hr during operation and 0.1 ml/kg/hr during postoperative 24 hours
  Other Names: normal saline
  Arms: control group

SUMMARY:
This study will be done to investigate perioperative lidocaine infusion on neutrophil extracellular trapping in the patients undergoing the robot-assisted prostatectomy.

DETAILED DESCRIPTION:
Neutrophil extracellular trapping by analyzing the meyloperoxidase, neutrophil elastase, citrullinated histone3

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled robot-assisted prostatectomy

Exclusion Criteria:

* lidocaine allergy Hx
* hemodynamic unstable patients
* weight < 40kg
* arrhythmia or bradycardia

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of citrullinated histone3 | 24 hours after surgery
  This will be obtained using ELISA.

SECONDARY OUTCOMES:
Concentration of meyloperoxidase | 24 hours after surgery
  This will be obtained using ELISA.
Concentration of neutrophil elastase | 24 hours after surgery
  This will be obtained using ELISA.

OTHER OUTCOMES:
the severity of postoperative pain using NRS | during postoperative 24 hours
  This will be measured using NRS (numeric rating scale; 0=no pain, 10=the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Young Eun Moon, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No